CLINICAL TRIAL: NCT04813198
Title: Feasibility and Preliminary Efficacy Testing of Therapy Integrating Peer-sharing, Technology, Aerobic and Resistance Training (TIPSTART) to Reduce Symptoms of Mental Illness in First-generation College Students
Brief Title: Feasibility of Therapy Integrating Peer-sharing, Technology, Aerobic and Resistance Training (TIPSTART)
Acronym: TIPSTART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Sean Mullen, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21184
Record Dates: First submitted 2021-03-20; First posted 2021-03-24 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Group Meetings
Keywords: mental health; exercise therapy; first-generation college students; academic stress; peer support; aerobic exercise; physical activity; depression; anxiety; resilience
MeSH Terms: conditions — Psychological Well-Being; Motor Activity; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention or a wait-list control condition.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI and co-Is will be blinded to group status. Survey and cognitive assessments will be delivered online without any reference to group. Interventionists have been trained to deliver program content but they are blinded to the primary outcomes of the study. Interviewers who gather qualitative data will be blinded to group status and primary outcomes of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIPSTART (Active Comparator): Following baseline testing, the study orientation and randomization, the TIPSTART group will engage in 5.5 hours (30 minutes, on 11 separate occasions, over 10 weeks) of training delivered through Zoom and supported by instructional and communication apps, and that is further supervised by our TIPSTART study navigators who will provide motivational support and detailed lifestyle behavioral prescriptions (150 to 300 minutes per week of aerobic and strength training, with mental practice of material discussed each week). Participants will also be asked to complete approximately 3 total hours of repeated testing that occurs online via surveys and face-to-face interviews for the 12-week study.
  Interventions: Behavioral: TIPSTART
- Wait-list Control (No Intervention): Following baseline testing, the study orientation and randomization, the wait-list control group will be asked to continue living life as usual until their delayed TIPSTART program is initiated. Participants will be asked to complete repeated online surveys and face-to-face interviews during the first 12 weeks, concurrently, with participants assigned to the TIPSTART intervention.

INTERVENTIONS:
Behavioral: TIPSTART — TIPSTART is a multimodal, cognitive behavior-based therapy integrating peer-sharing, technology, aerobic and resistance training.
  Arms: TIPSTART

SUMMARY:
The purpose of this randomized controlled clinical trial with first-generation college students with symptoms of mental illness is to test the preliminary feasibility and efficacy of TIPSTART, a multi-faceted, mental health and exercise training program-involving 5.5 hours of training delivered via assistance of remote technology, a licensed therapist and certified exercise behavior change specialist, and supported by peer pods-relative to a group receiving usual care. Students will confirm they are not currently treated with medication but have received mental health services in the past two years, and meet symptom cutoff criteria using a standard field screening assessment. It is hypothesized that the 10-week training program initiated at the onset of an academic semester will improve students' symptoms of anxiety and depression. Further, it is also expected that greater physical activity, self-efficacy, and social and academic engagement among participants in the TIPSTART group as compared to the usual care condition. Finally, the potential role of TIPSTART in changes in resilience, self-regulatory functioning and schoolwork-life balance will be explored.

DETAILED DESCRIPTION:
First-generation college students are at risk of serious mental illness. Relative to their peers, they are more likely to work full time, take fewer classes, use public transportation, and engage less with on-campus programs. Further, they report more traumatic stress, lower life satisfaction and less support from parents and peers. These findings are compounded by nationwide estimates of rising mental health issues across college campuses, where nontraditional students with financial hardship and/ or care-giving burdens represent the majority, and counseling services are increasingly under-resourced and overburdened. Moreover, less than 50% of college students are meeting public health guidelines for physical activity participation, a health behavior known to mitigate risk and enhance mental health.

Traditional four-year colleges and universities represent an opportunity to implement evidence-based mental health services, but many campuses are disconnected, low mental health-resource environments lacking well-coordinated programs specifically tailored for first-generation students, particularly cognitive behavior therapy (CBT) or programs guided by CBT principles, in concurrence with physical activity guidance and support. Evidence suggests that multimodal programs consisting of therapy integrating peer-support (in the form of pods), technology, aerobic plus resistance training (TIPSTART) has the potential to increase self-efficacy and self-regulatory strategies, utilization and maintenance of mental health services and behavior change techniques, and ultimately, reduce symptoms of mental illness. In the last decade, digital health interventions (e.g. smartphone apps) have been used with college-age populations to make therapy more accessible and exercise more enjoyable and socially-supported. App-based interventions have been successfully delivered as standalone interventions and have yielded positive effects on mental health outcomes, socio-emotional functioning and health behavior engagement.

The purpose of this randomized controlled clinical trial is to test the feasibility and preliminary efficacy and implementation of TIPSTART, a multi-faceted, mental health and exercise training program involving 5.5 hours of supervised training delivered via assistance of remote technology, a therapist and exercise behavior change specialist, and supported by peer pods (relative to a wait-list control group who will receive usual care) among first-generation college students with symptoms of mental illness. Students will confirm receipt of mental health services in the past two years, and meet cutoff criteria using a standard field screening assessment. It is hypothesized that the 10-week training program initiated at the onset of an academic semester will improve students' symptoms of anxiety and depression. Further, it is also expected that greater physical activity, self-efficacy, and social and academic engagement among participants in the TIPSTART group as compared to the usual care condition. Finally, the potential role of TIPSTART in changes in resilience, self-regulatory functioning and schoolwork-life balance will be explored.

ELIGIBILITY:
Inclusionary Criteria

* Enrolled at UIUC as a student with confirmed first-generation status (18 to 34 years old)
* Not currently taking medication for mental illness but have symptoms of mental illness and/or able to provide verifiable evidence of accessing mental health services in the past 2 years (proof of receipt of services is substitutable for record of diagnosis). Note: Should taking regular medication become necessary, participation in this study will in no way be impacted.
* Low-active (e.g., walk < two days/week, 20 minutes/day for last three months)
* English-speaking
* Not concurrently participating in another academic program, clinical trial or commercial program that may affect physical activity, diet, sleep, or meditation
* Not pregnant/lactating
* No pre-existing physical condition, recent injury or surgery that might be exacerbated by aerobic and resistive exercise
* Have smartphone (or willing to use portable device supplied by lab) and willing to install and use 'WellTrack' and 'Remind' apps and to allow researchers to pull data from apps (such as exercise entries and goals) and in-phone usage statistics of those apps at follow-up.

Exclusionary Criteria

* Not enrolled at UIUC as a student with first-generation status (18 to 34 years old)
* Taking medication for mental health condition or have no mental illness symptoms or unable to provide verifiable evidence of accessing mental health services in the past 2 years (proof of receipt of services is substitutable for record of diagnosis)
* Too active (e.g., walk > two days/week, >20 minutes/day for last three months)
* Not English-speaking
* Concurrently participating in another academic program, clinical trial or commercial program that may affect physical activity, diet, sleep, or meditation
* Pregnant/lactating
* Have pre-existing physical condition, recent injury or surgery that might be exacerbated by aerobic and resistive exercise
* Do not own smartphone (or are unwilling to use portable device supplied by lab) and/ or unwilling to install and use 'WellTrack' and 'Remind' apps and to allow researchers to pull data from apps and in-phone usage statistics of those apps at follow-up.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Anxiety | Change will be assessed from baseline to 12-week follow-up (assessed immediately post-intervention)
  The seven-item Generalized Anxiety Disorder (GAD-7) questionnaire will be used as our primary measure of anxiety. GAD-7 scores range from 0 (not at all) to 3 (nearly every day) and a composite score is computed by summing all responses. Scores range from 0 to 21 and will be recoded for ease of interpretation (higher scores will be interpreted as more favorable).
Depression | Change will be assessed from baseline to 12-week follow-up (assessed immediately post-intervention)
  The nine-item Patient Health Questionnaire (PHQ-9) will be used as our primary measures of depression. PHQ-9 scoring is identical to the GAD-7, however, the additional two items in increase the range from 0 to 27. Scores will be recoded for ease of interpretation (higher scores will be interpreted as more favorable).

SECONDARY OUTCOMES:
Feasibility and Implementation Evaluation | Assessed at week 6 and week 12 follow-up
  One-hour interviews were conducted with a sub-sample of participants. Specifically, participants were asked open-ended about aspects of their life (financial, emotional, familial, social, health) they felt were most impacted by their experiences in the TIPSTART program, as well as the most memorable/standout services. In addition, participants were asked about any negative or unintended consequences of their participation, such as deterioration of symptoms, adverse events, novel symptoms, unwanted events, etc.
Intervention adherence | Assessed across the 10-week intervention
  The percentage of sessions attended out of 10, as well as the percentage of total weeks participants reported adherence to the minimum physical activity prescription (public health guidelines of 150 minutes) and weekly mental exercises, will be used to represent adherence to our TIPSTART intervention.
Knowledge of mental health services and resources | Assessed at baseline, week 6 and week 12 follow-up
  Participants were asked to indicate (by checking boxes), "Which of the following on-campus/ remote mental health resources at your university are you aware of (whether or not you have utilized them). Please check all that apply."
Utilization of mental health services | Assessed at baseline, week 6 and week 12 follow-up
  Please describe any in-person or remote mental health resources you have utilized (not affiliated with your university) over the past 5 weeks. This could include, but is not limited to in-person talk therapy or telecounseling with a private practice therapist, a rehabilitation center, outpatient clinic, app-based services, etc. Which of the following on-campus/ remote mental health resources at UIUC have you used in the past 5 weeks? Which of the follow on-campus/ remote mental health resources at UIUC have you used the most in the past 5 weeks? (if you have not used any, please select "None"). How many times have you used this resource in the past 5 weeks?
Self-reported leisure-time exercise | Assessed at baseline, week 6 and week 12 follow-up
  Physical activity at baseline will be assessed via the Godin-Shephard Leisure-Time Physical Activity Questionnaire (GLTEQ; Godin, 2011). The GLTEQ assesses leisure-time activity across three modes of activity: strenuous, moderate, and mild, in terms of frequency and duration. Weekly frequencies of strenuous, moderate, and mild activities were multiplied by nine, five, and three, respectively to create the total score or number of units. According to this score, 24 units or more is indicative of an active individual, whereas any score below 24 is indicative of a non-active individual.
Process of Recovery | Assessed at baseline, week 6 and week 12 follow-up
  The 15-item Questionnaire about the Process of Recovery (QPR) will be used to assess meaningful aspects of recovery. Each item is scored on a 4-point scale (0= disagree strongly, 1=disagree, 2=neither agree nor disagree, 3=agree, 4=agree strongly) and items are summed to create a composite. Higher scores are indicative of recovery.
Resilience | Assessed at baseline, week 6 and week 12 follow-up
  The 17-item Adult Resilience Measured-Revised (ARM-R; Jeffries, McGarrigle, & Ungar, 2018) will be used to assess perceived social-ecological resilience. The ARM-R utilizes a 5-point Likert scale (ranging from 1=Not at all to 5=A lot) and it has two subscales: personal (10 items) and relational (7 items) resilience. Items are summed creating minimum and maximum scores of 10 to 50 for personal resilience and 10 to 35 for relational resilience, where higher scores reflect higher resilience.
Perceptions of Academic Stress | Assessed at baseline, week 6 and week 12 follow-up
  The 18-item Perceptions of Academic Stress (PAS) scale by Bedewy and Gabriel (2015) was used to assess academic domain-specific stress. For example, participants are asked to indicate the extent to which they agree with statement such as, "Am confident that I will be a successful student," on a 5-point Likert scale (1=Strongly disagree, 5=Strongly agree). The PAS scale also addresses sources of stress, such as, "Teachers have unrealistic expectations of me" (1=Strongly agree, 5=Strongly disagree). Subscale scores will be computed by summing respective items and calculating an un-weighted averaged. Some scores will be reversed to ensure that lower composite scores reflect lower perceived stress.
Academic Engagement | Assessed at baseline, week 6 and week 12 follow-up
  Academic engagement was assessed via self-report using a 4-item questionnaire by Hu and Wolniak (2013). Specifically, participants were asked to indicate the frequency they they worked with other students on schoolwork outside of class, discussed readings or classes with students and faculty outside of class, and worked harder than thought to meet an instructor's expectations on a 6-point Likert scale (response options ranged from 1=less than once a month to 6=four or more times a week). Items are summed and averaged and higher scores indicate higher levels of academic engagement.
Social Engagement | Assessed at baseline, week 6 and week 12 follow-up
  Social engagement was assessed via self-report using a scale by Hu and Wolniak (2013). Specifically, participants were asked to indicate the frequency they they participate in events sponsored by a fraternity or sorority, residence hall activities, events by groups reflecting own culture heritage, and community service activities on a 5-point Likert scale (response options ranged from 1=never to 5=very often). Items are summed and averaged and higher scores indicate higher levels of academic engagement.
Schoolwork life-balance | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Six items (e.g. "Because of my school work, I have no time," "I have enough time for my friends") were used to assess perceived time availability for school and social life. Items were rated on a 6-point Likert ranging from "Completely Disagree" to "Completely Agree." Items 2 and 3 are reverse-coded. A composite score is derived by adding and averaging, with higher scores reflecting greater balance between schoolwork and life.
Self-efficacy to regulate school-life | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  The Self-efficacy to Regulate Work and Life Questionnaire is a 5-item questionnaire that assesses how confident individuals are in regulating their work and non-work domains (Chan et al., 2016).The five items include: 1) "How confident are you in changing your lifestyle to achieve a good work-life balance?," 2) "How confident are you in finding out how to balance work and life?," 3) "How confident are you in achieving your ideal work-life balance?," 4) "How confident are you in implementing strategies to achieve work-life balance?," and 5) "How confident are you in inventing ways to balance your work and life?." Responses to all items are based on a scale ranging from 0 (cannot do at all) to 100 (highly certain can do). The composite score is calculated by summing and averaging the five items, with higher scores indicating that individuals are more confident in their abilities to cope with work-life challenges.
Physical activity self-regulation | Assessed at baseline, week 6 and week 12 follow-up
  The Physical Activity Self-Regulation Scale (PASR-12; Umstattd, Motl, Wilcox, Saunders, & Watford, 2009) will be used to assess the use of self-regulation strategies for engaging in physical activity. The PASR-12 is a 12-item questionnaire with responses ranging from 1 (never) to 5 (very often). A total score can be calculated by summing up responses to all the items. There are also six subscales (self-monitoring, goal-setting, social support, reinforcement, time management, and relapse prevention), however, research by our lab has found that this scale is not uni-dimensional. We will use a modified version of the scale. Higher score reflects higher use of self-regulation strategies.
Exercise-related planning | Assessed at baseline, week 6 and week 12 follow-up
  The Exercise Planning and Schedule Scale (EPSS; Rovniak, Anderson, Winett, & Stephens, 2002) is a 10-item questionnaire that assesses exercise scheduling and planning. Each question is based on a 5-point Likert scale, ranging from 1 (does not describe me) to 5 (describes me completely). The EPSS composite score is calculated by reverse-scoring items 2, 3, and 7 then summing and averaging the 10-items to create a composite score. Higher scores indicate more scheduling and planning done for exercise. In addition, we used a novel questionnaire asking participants the extent to which the following 5 statements are true (4-point Likert scale range: 1=Not at all true, 4 = Absolutely true). "For the next month, I have already planned... which days (frequency; F), the intensity (I), how long (time; T), which types (T), and where (location; L) I will exercise." F.I.T.T.L. scores will be averaged and higher scores represent greater planning.
Self-efficacy to overcome barriers to exercise | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  A 13-item questionnaire will be used to assess self-efficacy specific to possible barriers affecting exercise adherence. All items will be answered on a 0-100% Likert scale in increments of 10%. Prior research suggests that this may not be a uni-dimensional scale and therefore a composite will be based on a 4-item composite. These four items best reflect participants' confidence to self-regulate in the face of actual barriers, including exercising regularly in the face of bad weather, while on vacation, without encouragement, and when under personal stress. These four items will be averaged to generate our main outcome of interest, and the remaining nine items will be assessed for exploratory purposes.
Self-efficacy for lifestyle physical activity | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Self-efficacy to engage in physical activity will be assessed using the Lifestyle Self-efficacy Scale (E McAuley et al., 2009), which asks participants about their belief in their ability to be physically active five or more times per week at a moderate intensity, for at least 30 minutes, for six months.
Social support for exercise | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Participants were asked to indicate the frequency (0=Never, 4=Very Often) that they received companionship, informational, and esteem support from friends or an expert (6 total sub-scales derived from the Multidimensional Social Support Scale; Chogahara, 1999). Each 5-item sub-scale score will be computed by summing and averaging the five numeric responses. Higher scores reflect higher levels of perceived social support.

OTHER OUTCOMES:
Demographics | Assessed at baseline
  Age, gender, year in college, first-generation status (mother's & father's highest educational degree), race, ethnicity, and employment status will be assessed for descriptive purposes.
Grade-point average | Assessed at baseline and week 12 follow-up.
  Student grade-point average and registered course hours will be assessed via self-report to gauge how well students are doing academically.
Perceived height and weight | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Two items assessing self-reported height and weight will be used to calculated body mass index.
Economic hardship | Assessed at baseline
  Four items were used to assess economic hardship. One item assessed the number of hours per week to cover basic necessities (ranging from 1-5 hours/week to 16+ hours), and three items ask the extent respondents agree with specific statements. For example, "The time I spend earning money to cover my basic necessities (including tuition) frequently takes away from the time I have to study." The three statements are rated on a Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree).
College shock | Assessed at baseline
  Difficulty with transitioning to college or "college shock" was assessed via two items. Specifically, "My transition to college has been smooth" (1=strongly agree to 5=strongly disagree) and "Which statement best explains your previous educational experience? My previous educational experience..." (1=completely prepared me for my university's rigor; 4=has not at all prepared me for my university's rigor). Lower scores indicate less college shock.
Medication use | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Participants were initially excluded from the trial if they were already taking medication, but it was not ethical to subsequently remove participants if they later required medication for mental illness (or other conditions) upon commencement of the study. We therefore asked, "Are you currently diagnosed with a condition that requires daily or weekly prescription medication (yes/no)?" For those who began taking medication, we also asked, "In the past month, how often did you take your medications as the doctor prescribed?" (1=Less than half the time, 5=All of the time).
Caffeine use | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Consumption of caffeinated beverages (soft drinks, tea, coffee) was assessed via single self-reported item with five response options ranging from "None" to "More than 8 cups/day."
Alcohol use | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Consumption of alcohol was assessed with a single item with nine response options ranging from "None" to "4 or more drinks per day/week, otherwise 0-1 drinks/day." In addition, we assessed participants "Do you drink alcohol in moderation, according to the guidelines set forth by the American Heart Association (i.e. 1-2 drinks per day for men and 1 drink per day for women)? Yes or No.
Smoking behavior | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Smoking behavior was assessed via self-report (Ciccolo et al., 2014). Participants were asked whether or not "even a puff" was taken within the last 7 days, 24 h, and the date of the last puff. This allows for an examination of the number of smoking cessation outcomes, including initial abstinence (24-h abstinence), time to first lapse (first smoking event following initial abstinence), time to relapse (smoking at least 5 cigarettes/day for 3 consecutive days), and prolonged abstinence.
Health status | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  A single item, "How would you rate your overall health status" (1=Poor, 5=Excellent) was used as an overall index of health status.
Perceived Stress | Assessed at baseline, week 6 and week 12 follow-up
  The Perceived Stress Scale (PSS), developed by Cohen, Kamarck, and Mermelstein (1983) will be used to measure perceived psychosocial stress. The PSS is a 10-item scale that measures the extent to which situations are perceived as stressful. Responses range from 0 (Never) to 4 (Very often) and higher scores indicate a higher level of perceived stress. The Brief Job Stress Questionnaire, developed by Kawada and Otsuka (2011), is a 15-item scale measuring job stress. It focuses on the evaluation of job demands, job control, job support, and degree of job satisfaction. Responses range from 1 (Agree) to 4 (Disagree) and higher scores indicate a lower level of stress.
Exercise self-efficacy | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Participants' beliefs in their ability to continue exercising in the future was assessed via McAuley's (1993) 6-item Exercise Self-Efficacy scale. Respondents rate their confidence to carryout exercise for the next six months, three times per week at a moderate intensity, for 40+ minutes per session. The scale is comprised of a 100-point percentage scale using 10-point increments, ranging from 0% (not at all confident) to 100% (highly confident). Total scores are calculated by averaging all six item responses where higher scores indicate higher self-efficacy.
Exercise self-schema | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  The Exercise Self-Schema Questionnaire (ESSQ; Kendzierski, 1988) will be used to assess participant "self-definition" or identity as an exerciser. The ESSQ was originally a 9-item scale and we are using a modified version which includes an additional item reflecting self-certainty ratings for each self-description item, as well as an extra question reflecting self-description, -importance, and -certainty with regard to "I am someone who will always be an exerciser" (Mullen, 2011). This 12-item version of ESSQ utilizes the same 11-point Likert Scale, ranging from 1 (does not describe me) to 11 (describes me). Items representing each subscale (self-description, importance, certainty) will be averages with higher scores indicating higher levels of each aspect of self-as-exerciser identity. Exerciser schematics will also be determined by categorizing responses to self-description and importance items that fall within the 8 to 11 range.
Eating identity | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  The Healthy Eating Self-Schema Questionnaire (Kendzierski & Costello, 2004) was used to assess participants' identity in relation to food. Specifically, self-descriptiveness of each of three key phrases, i.e., "healthy eater," "someone who eats in a nutritious manner," and "someone who is careful about what I eat," are self-rated on an 11-point scale ranging from 1 (does nor describe me) to 11 (describes me). Participants also rated importance of the phrases "to the image you have of yourself regardless of whether or not you are someone who is ..." Importance ratings are from 1 (not at all important) to 11 (very important). Participants are classified as healthy eater schematics if they rate at least two of the three descriptors as very self-descriptive (ratings of 8-11) and rated at least two of the three descriptors as very important to their self-image (ratings of 8-11).
Exercise-related outcome expectations | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Participants' expectations about the outcomes of this intervention will be assessed using the Multidimensional Outcome Expectancies for Exercise Scale (MOEES). It is a 15-item questionnaire measuring physical outcome expectancies, social outcome expectancies, and self-evaluative outcome expectancies. Responses range from 1 (strongly disagree) to 5 (strongly agree). The total score for each subscale is calculated by summing the items, with higher scores being indicative of higher outcome expectations for exercise.
Anticipated negative affect related to exercise | Assessed at baseline, week 6 and week 12 follow-up
  Anticipated negative emotions will be assessed via the Anticipated Negative Affect Questionnaire (ANAQ; Wang, 2011). The ANAQ asks participants to anticipate how they may feel not regularly participating in physical activity. The ANAQ consists of 5 bi-polar items: "relaxed/tense," "not guilty/guilty," "no regret/regret," "not angry/angry," and "displeased/pleased." The ANAQ scale ranges from 1 to 7. Anticipated negative affect is scored based upon the number provided for each individual question, with higher scores indicating more negative emotions.
Exercise motivation | Assessed at baseline, week 6 and week 12 follow-up
  The Exercise Motivations Inventory-2 was used to assess the type of reasons one has for participating in an exercise program (and their relative strength). Only three of the 14 total sub-scales were implemented. Specifically, four items assessing appearance, three items assessing positive health, and four items assessing affiliation were used. Composite scores will be computed for each sub-scale by summing and averaging the numeric responses from the 6-point Likert-scale (ranging from 0=Not at all true for me, 5=Very true for me). Higher sub-scale scores reflect strong motivation for the respective reason for exercising.
Sleep quality | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  The Pittsburgh Sleep Quality Index (PSQI; Buysse et al 1989) is composed of 19 self-rated questions and 5 questions rated by a bed partner or roommate (only the self-rated items are used in scoring the scale). The self-administered scale contains 15 multiple-choice items that inquire about frequency of sleep disturbances and subjective sleep quality and 4 write-in items that inquire about typical bedtime, wake-up time, sleep latency, and sleep duration. The 5 bed partner questions are multiple-choice ratings of sleep disturbance.
Frequency of forgetting | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  The general rating of memory (first item) subscale was used from the Frequency of Forgetting scale (Zelinski & Gilewski, 2004). Specifically, respondents were asked, "How would you rate your memory in terms of the kind of problems that you have?" where 1=Major Problems and 7=Major Problems. Higher scores indicate more memory problems.
Memory strategies | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  The 20-item Strategies subscale of the Meta-memory Questionnaire (Troyer & Rich, 2002) was used to assess the extent to which participants' engaged in cognitive and behavioral strategies aimed at improving their memory over the past 2 weeks. Responses are rated on a 5-point Likert scale ranging from 0 (Never) to 4 (All the time). Items are summed and higher scores represent higher usage of memory aids and strategies.
Exercise-specific memory self-efficacy | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Self-efficacy for remembering certain aspects of starting a new exercise program (e.g. public health recommendations, correct movements/form, optional modifications, and how to evaluate progress) was assessed with a novel questionnaire by Mullen and his colleagues. Responses ranged from 0% (Not at all confident) to 100% Completely confident). Composite scores are calculated by averaging the four-item sub-scales targeting self-efficacy for remembering the aforementioned aspects of aerobic, strength, and flexibility training. Higher scores indicate greater confidence in memory for each aspect of exercise training.
Exercise Experience | Assessed at baseline
  Lifelong exerience with structure exercise. For example, "Over the course of your lifetime, overall, how much experience do you have doing structured exercise within a fitness facility that included some combination of aerobic, strength, and flexibility training? (ONLY include years when you exercised at a facility for 6+ months on a regular basis)."
Fitness Technology Experience | Assessed at baseline
  Lifelong experience playing exergames and using smartphone apps to improve health and fitness, and to brain-train, was assessed.
Future time perspective | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  The Future Time Perspective (FTP; Lang & Carstensen, 1994) scale includes 10 items answered by indicating agreement on a 7-point Likert-type scale (from 1= very untrue, to 7 = very true). The last three items of the FTP scale are reverse-coded. The total score is based on an un-weighted averaged of all 10 items. Higher scores reflect the perspective of a longer time horizon.
Mindfulness | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  Mindfulness will be assessed via the Mindfulness and Attention Awareness Scale (MAAS; Brown & Ryan, 2003). The MAAS is a 15-item measure of dispositional mindfulness in the context of day to day activities. Participants use a Likert-type response scale ranging from 1 (almost always) to 6 (almost never). The total score is calculated by summing the response to all items, and higher scores reflect a higher level of dispositional mindfulness.
Grit | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  The original 12-item of the Grit scale (Duckworth et al, 2007) was used to assess the trait-level personality construct known as "grit." However, the shorter version (Grit-S; Duckworth & Quinn, 2009) will be derived from the larger scale, to be used in the calculation of total scores, given its superior psychometric properties. Higher scores will indicate higher levels grittiness.
Personality dimensions | Assessed at baseline, week 6 and week 12 follow-up (assessed immediately post-intervention)
  The 44-item Big Five Inventory (John, Donahue, & Kentle, 1991) was used to assess the personality dimensions of Extraversion, Agreeableness, Conscientiousness, Neuroticism, and Openness to experience. Respondents are asked to consider the statement, "I see myself as someone who..." and then rate the extent to which they agree with a list of traits on a scale from 1 (Disagree Strongly) to 5 (Agree Strongly). Each subscale's items are summed and averaged. Higher scores reflect higher levels of personality dimension.
Sitting time | Assessed at baseline, week 6 and week 12 follow-up
  Sitting time was measured via self-report, for weekdays and weekends, using the Sitting Time Questionnaire (Marshall et al, 2010). Participants are asked to, "Please estimate how many hours you spend sitting each day, an the following situations, including while traveling to and from places, while at work, while watching television, while using a computer at home, and for all other leisure time, not including television." Each category is summed and averaged across weekdays and weekends, separately.
Active choices | Assessed at baseline, week 6 and week 12 follow-up
  The English-translated version of the Activity Choice Index (Mullen et al, 2016) was used to assess deliberate substitution of more effortful choices to engage in lifestyle physical activity. Specifically, self-reported lifestyle physical activities typical of the previous month were assessed with six items (using stairs or escalators, walking instead of using transportation, parking away from one's destination, using work breaks to be physically active, choosing to stand up instead of sitting, and choosing hand work instead of mechanic/automatic). Items are rated on a 5-point Likert scale (i.e., 1 = never, 5 = always). The composite score is calculated by averaging an un-weighted sum of each item.
Cardiorespiratory fitness | Assessed at baseline, week 6 and week 12 follow-up
  Cardiorespiratory fitness (CRF; Jurca et al. 2005) will be estimated according to an established algorithm involving gender, age, body mass index, resting heart rate, and a unique self-reported physical activity (SRPA) measure. The SRPA is a single exercise history question in which participants are asked to identify one of five physical activity categories that reflect their usual pattern of daily physical activity including activities associated with home and family care, transportation, work, exercise and wellness, and leisure or recreation. Given that the study design is entirely remote, resting heart rate will be assessed via open-ended response during survey administration using a 60-sec instructional video.
Adverse and unintended events | Assessed weekly during intervention sessions
  Study navigators will ask participants if they have experienced any adverse or unintended consequences as function of the intervention. They will also monitor electronic correspondence and any reports of injury or related events.
Intentions | Assessed at baseline, week 6 and week 12 follow-up
  Per the recommendations of Leon et al (2007) for reducing bias from dropout within randomized controlled trials, we assessed intent to dropout and related questions. Specifically, five items will be used to assess intentions to adhere to the TIPSTART program and comply with our study assessments (How likely is it that you will complete the next survey?), complete the study (How likely is it that you will complete the entire study?), and behavioral prescriptions associated with the intervention (If you are assigned to receive TIPSTART, how likely is it that you will adhere to our 10-week program? How likely is it that you will adhere to the exercise prescription [achieving 150-300 minutes of moderate intensity physical activity per week] for the duration of the study? How likely is it that you will complete our weekly online mental health sessions and remote check-ins?). Participants are asked to respond on a 0 to 9 Likert scale that ranges from "Not at all" (0) to "Extremely" (8).
Attention checks | Assessed at baseline, week 6 and week 12 follow-up
  Four items will be used to ensure that participants are fully engaged and respond to the survey questions to the best of their ability. Items will be spaced throughout the survey (for example, participants will be asked to "Please select the number 3 among the responses below"). Each item will be assessed for accuracy and an average will be computed based on all four responses.

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Mullen, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Louise Freer Hall, Exercise Technology & Cognition Laboratory, Rooms 284-284A, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Mullen S, Luo Y, Adamek J, Phansikar M, Mackenzie M, Roberts B, Larrison CR. Path Analysis of Effects of First-Generation Status on Physical Activity and 4-Year College Degree Completion. J Evid Based Soc Work (2019). 2024 Jan 2;21(1):104-116. doi: 10.1080/26408066.2023.2265922. Epub 2024 Jan 3. PMID 37811659
- See also: University of Illinois students interested in determining their study eligibility should contact us using this web form. — http://exercisestudy.com/tipstart